CLINICAL TRIAL: NCT02172157
Title: Investigation of the Metabolism and Pharmacokinetics of 20 μg (Calculated as Free Base) [14C]BI 1744 CL Administered as a 3-hour Infusion and 40 μg (Calculated as Free Base) [14C]BI 1744 CL Administered as an Oral Solution.
Brief Title: Investigation of the Metabolism and Pharmacokinetics of [14C]BI 1744 CL and [14C]BI 1744 CL Administered as an Oral Solution in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1222.9
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — olodaterol

ARMS (2):
- BI 1744 CL i.v. (intravenous) infusion (Experimental)
  Interventions: Drug: BI 1744 CL i.v.
- BI 1744 CL Oral solution (Active Comparator)
  Interventions: Drug: BI 1744 CL oral

INTERVENTIONS:
Drug: BI 1744 CL i.v.
  Arms: BI 1744 CL i.v. (intravenous) infusion
Drug: BI 1744 CL oral
  Arms: BI 1744 CL Oral solution

SUMMARY:
Primary objective:

To determine the basic pharmacokinetics of BI 1744 BS, its metabolite BI 1744 BS - glucuronide and [14C]-radioactivity including excretion mass balance, excretion pathways and metabolism following intravenous and oral administration of [14C]BI 1744 CL

Secondary objective:

To determine safety and tolerability following intravenous and oral administration of [14C]BI 1744 CL in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
* Age ≥18 and ≤45 years
* Body mass index (BMI) ≥18.0 and BMI ≤30.0 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic, or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to study drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration until after the last sample from Visit 2 is collected
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking during the stay in the trial centre
* Alcohol abuse (more than on average 2 units of alcoholic beverages per day or more than 14 units per week (1 unit equals 1 pint [285 mL] of beer or lager, 1 glass [125 mL] of wine, 25 mL shot of 40% spirit))
* Drug abuse
* Blood donation (more than 100 mL within 60 days prior to study drug administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial until follow-up examination)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of study centre
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)

Exclusion criteria specific for this study:

* Veins unsuitable for infusion and blood sampling
* PR interval >220 ms or QRS interval >120 ms
* Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton (excluding spinal column)), during work or during participation in a medical trial in the previous year
* Irregular defecation pattern (less than once per 2 days)

The following exclusion criteria are specific for this study due to the known class side effect profile of β2-mimetics:

* Asthma or history of pulmonary hyperreactivity
* Hyperthyrosis
* Allergic rhinitis in need of treatment
* Clinically relevant cardiac arrhythmia
* Paroxysmal tachycardia (>100 beats per minute)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Individual time course profiles of [14C]-radioactivity in whole blood, plasma, urine and faeces | Pre-dose and up to 216 hours after start of drug administration
Individual time course profiles of of the analyte in plasma and urine | Pre-dose and up to 216 hours after start of drug administration
Rate and extent of excretion mass balance based on the total radioactivity in urine and faeces | Pre-dose and up to 216 hours after start of drug administration
C (concentration) blood cells/C plasma ratio of [14C] -radioactivity | Pre-dose and up to 96 hours after start of drug administration
Plasma and urinary concentrations of the analyte | Pre-dose and up to 216 hours after start of drug administration
Whole blood, plasma and urinary concentrations of the [14C]-radioactivity | Pre-dose and up to 216 hours after start of drug administration
Cmax (maximum concentration of the analyte(s) in plasma) | Up to 96 hours after start of drug administration
tmax (time from dosing to the maximum concentration of the analyte(s) in plasma) | Up to 96 hours after start of drug administration
AUC (area under the concentration-time curve at different time points) | Up to 96 hours after start of drug administration
λz (terminal rate constant in plasma) | Up to 96 hours after start of drug administration
t1/2 (terminal half-life of the analyte(s) in plasma) | Up to 96 hours after start of drug administration
MRTpo and MRT, respectively (mean residence time of the analyte(s) in the body after po and iv administration) | Up to 96 hours after start of drug administration
CL and CL/F (total clearance of the analyte in plasma after iv and oral administration) | Up to 96 hours after start of drug administration
Vz and Vz/F (apparent volume of distribution during the terminal phase λz following an iv and oral dose) | Up to 96 hours after start of drug administration
Vss (apparent volume of distribution at steady state following intravascular administration) | Up to 96 hours after start of drug administration
Ae0-tz (amount of analyte that is eliminated in urine within the time interval zero to tz) | Up to 216 hours after start of drug administration
fe0-tz (fraction of analyte excreted in urine within the time interval zero to tz in % of dose) | Up to 216 hours after start of drug administration
Aefaeces,0-tz (amount of analyte excreted in faeces within the time interval zero to tz) | Up to 216 hours after start of drug administration
fefaeces,0-tz (fraction of analyte excreted in faeces within the time interval zero to tz in % of dose) | Up to 216 hours after start of drug administration
CLR,t1-t2 (renal clearance of analyte from the within the time interval t1 to t2) | Up to 216 hours after start of drug administration
Fa (fraction of drug absorbed after oral administration) based on total radioactivity data after oral and iv administrations | Up to 216 hours after start of drug administartion
F (oral bioavailability) based on parent BI 1744 CL concentration data after oral and iv administration | Up to 216 hours after start of drug administartion

SECONDARY OUTCOMES:
Number of patients with clinical significant changes in vital signs | Baseline and up to 24 days after drug administration
Number of patients with abnormal findings in physical examination | Baseline and up to 24 days after drug administration
Number of patients with clinical significant changes in 12-lead ECG (electrocardiogram) | Baseline and up to 24 days after drug administration
Number of patients with changes in Telemetry (iv treatment only) | -0.5 and up to 24 h after iv drug administration
Number of patients with abnormal changes in laboratory parameters | Baseline and up to 24 days after drug administration
Number of patients with changes in Bedside potassium monitoring (iv treatment only) | Pre dose and up to 3.5 hours after drug administration
Number of patients with adverse events | Up to 24 days after drug administration
Assessment of tolerability (global tolerability (both treatments) and local tolerability (iv treatment only)) on a 4 point scale | At discharge on day 10